CLINICAL TRIAL: NCT06890221
Title: Impact of PErioperative Nutrition Intervention on Bioimpedance Phase Angle (IPENIPA) In Breast Cancer Patients: A Double-Blinded Randomized Controlled Trial
Brief Title: Impact of PErioperative Nutrition Intervention on Bioimpedance Phase Angle (IPENIPA) In Breast Cancer Patients
Acronym: IPENIPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Collaborators: B-Crobes Laboratory (M) Sdn Bhd (Unknown)
Responsible Party: Principal Investigator, Soo Wai Yin, Medical Doctor, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IPENIPA; MECID 2024521-13747 (Other: Universiti Malaya); NMRR ID-24-01805-DNE (Other: National Medical Research Register (Malaysia))
Record Dates: First submitted 2025-03-16; First posted 2025-03-21 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3); Mastectomy Patient
Keywords: bioimpedance phase angle; nutritional intervention; oral nutritional supplement

STUDY DESIGN:
Intervention Model Description: Double blinded
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo
- Cohort B (Active Comparator): Oral nutrition supplement
  Interventions: Dietary Supplement: B-Crobes intake complete nutrition

INTERVENTIONS:
Dietary Supplement: B-Crobes intake complete nutrition — Contains whey and plant based proteins, enriched with prebiotics and probiotics, Ca-Hmb, minerals and multivitamins.
  Other Names: Oral nutrition supplement
  Arms: Cohort B
Dietary Supplement: Placebo — Contains full cream dairy milk
  Arms: Cohort A

SUMMARY:
The goal of this clinical trial is to measure the mean difference of phase angle after nutritional intervention in breast cancer patients. The main question it aims to answer is:

1. Can perioperative nutrition interventions improve phase angle in relation to other bioimpedance parameters, handgrip strength and surgical outcomes in breast cancer population?

Researchers will compare oral nutritional supplement to a placebo to see if oral nutritional supplement can improve phase angle.

Participants will:

1. Be randomized into either arm
2. Take oral nutritional supplement or placebo according to the result of randomization for 7 days preoperatively and 30 days postoperatively
3. Have their measurements (weight, height, phase angle, handgrip strength) done at least 7 days preoperative, 1 day preoperative and 30 days postoperative

ELIGIBILITY:
Inclusion Criteria:

* Female
* Histopathologically confirmed operable breast cancer
* Aged 18 of years and above
* Consented and scheduled for mastectomy

Exclusion Criteria:

* On enteral supplementation prior to the study
* Lactose intolerance
* Pregnant or lactating
* Previous history of gastrectomy or small bowel resection surgery
* Advanced breast cancer staging, presence of pacemaker, decompensated liver disease, end stage renal failure, uncontrolled diabetes, on steroid therapy or complementary traditional medications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 114 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean difference of phase angle after nutritional intervention | From enrollment to 30 days post operation
  To measure the mean difference of phase angle between groups after nutritional intervention

SECONDARY OUTCOMES:
Changes in handgrip strength | From enrollment to 30 days post operation
  To study the changes on handgrip strength, body composition by bioimpedance analysis (skeletal muscle mass, skeletal muscle mass index, fat free mass and fat mass) after nutritional interventions.
Correlation of phase angle with bioimpedance analysis parameters | From enrollment to 30 days post operation
  To describe the correlation of phase angle with nutritional status, handgrip strength, and body compositions by bioimpedance analysis (Skeletal muscle mass, skeletal muscle mass index, fat free mass, and fat mass).
Potential factors associated with postoperative complications | From enrollment to 30 days post operation
  To identify the potential factors associated with complications and readmission in 30-days post-mastectomy participants.
Cutoff value of phase angle | From enrollment to 30 days post operation
  To identify the cutoff value of PA in relation to GLIM malnutrition, nutrition risk, and sarcopenia

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Malaya Medical Centre, Petaling Jaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided